CLINICAL TRIAL: NCT04498156
Title: Awareness of Diagnosis and Treatment of Chronic Kidney Disease in Patients With Type 2 Diabetes
Brief Title: Survey of Patient and Physician Awareness and Values to the Diagnosis and Treatment of Reduced Kidney Function (Chronic Kidney Disease) in Patients With High Blood Sugar Level (Type 2 Diabetes) (AWARE-CKD in T2D)
Acronym: AWARE-CKD
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: LMC Diabetes & Endocrinology (Unknown)
Responsible Party: Sponsor
Other Study IDs: 21225
Record Dates: First submitted 2020-07-31; First posted 2020-08-04 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Renal Insufficiency, Chronic
Keywords: Chronic kidney disease (CKD); Type 2 Diabetes (T2D); Patient awareness; Physician awareness; Interaction patient physician
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CKD-Patients: Cohort consisting of adult patients with a known diagnosis of type 2 diabetes and evidence of chronic kidney disease (CKD)
  Interventions: Other: No intervention
- Physicians treating CKD: Cohort consisting of licensed general practitioners, endocrinologists and nephrologists who are currently treating patients with both chronic kidney disease (CKD) and type 2 diabetes
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention, observational study

SUMMARY:
In this survey study, researchers want to find out more about how physicians are treating patients diagnosed with reduced kidney function (chronic kidney disease, CKD) and high blood sugar level (type 2 diabetes); what physicians know about the different treatment options available; and how they use this knowledge to treat their patients successfully. Additionally, researchers want to gather information about patient's awareness of their disease and which criteria they consider important for their treatment of the disease.

The study will survey a total of 150 patients with type 2 diabetes: 50 patients with mild CKD; 50 patients with moderate CKD; and 50 patients with severe CKD. Patients eligible for this study can be male or female and should be at least 18 years old. In addition, a total of 150 physicians will be surveyed. Physicians eligible for this study may be general practitioners, endocrinologist, or nephrologists.

DETAILED DESCRIPTION:
The primary objective in this study is to assess the awareness, values and preferences of patients and physicians with respect to the risks, consequences and management of chronic kidney disease (CKD) in patients with type 2 diabetes.

Secondary objectives aim to assess awareness of available CKD treatments, referral tools and communication between patients and physicians.

Both patients and physicians will complete a survey that consists of various questions regarding the knowledge of disease, values and treatments, patient-physician interaction, physician referral tools and disease risk management.

ELIGIBILITY:
Inclusion Criteria:

* For patient cohort:

  * Diagnosis of type 2 diabetes
  * eGFR < 60 ml/min per 1.73 m2 (measured within the last year) OR eGFR ≥ 60 ml/min per 1.73 m2 and uACR ≥ 2 (measured within the last year)
  * No documented non-diabetic etiology for renal disease
* For physician cohort:

  * Licensed general practitioner, endocrinologist or nephrologist
  * Currently providing care for patients with chronic kidney disease and type 2 diabetes

Exclusion Criteria:

* Patients with chronic kidney disease and type 2 diabetes who are physicians
* Physicians with chronic kidney disease and type 2 diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with CKD and T2DM and treating general practitioners, endocrinologists, nephrologists in Canada
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Awareness of chronic kidney disease in T2D | 1 day
  Awareness will be summarized descriptively based on various survey questions.
Values regarding chronic kidney disease in T2D | 1 day
  Values regarding risks, consequences and management of chronic kidney disease will be summarized descriptively based on various survey questions.
Preferences regarding chronic kidney disease in T2D | 1 day
  Preferences regarding risks, consequences and management of chronic kidney disease will be summarized descriptively based on various survey questions.

SECONDARY OUTCOMES:
Awareness of available treatments for chronic kidney disease in T2D | 1 day
  Awareness of available treatments will be summarized descriptively based on various survey questions.
Physician awareness of available referral tools for the management of chronic kidney disease in T2D | 1 day
  Physician cohort only. Referral tools may comprise of various standard guidelines (e.g. KidneyWise, KDIGO guidelines, Diabetes Canada guidelines). A higher number of referral tools known by physicians indicates a better awareness of CKD referral tools.
Time point of communicated CKD diagnosis | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Many Facilities, Multiple Locations, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.